CLINICAL TRIAL: NCT01849432
Title: Probing Amygdalo-Cortical Circuitry in Anxiety Disorders
Brief Title: Study of Brain Circuitry in Anxiety Disorders
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Rauch, President, Psychiatrist in Chief, Mclean Hospital
Other Study IDs: 1R01MH070730-01A2 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Posttraumatic Stress Disorder; Panic Disorder; Specific Phobias
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Panic Disorder; Phobia, Specific

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Healthy Controls
- Posttraumatic Stress Disorder: Participants with Posttraumatic Stress Disorder
- Panic Disorder: Participants with Panic Disorder
- Specific Phobia: Participants who have specific phobias

SUMMARY:
A diverse body of research has implicated the amygdalo-cortical circuitry in the pathophysiology of anxiety disorders. For example, one model of PTSD posits exaggerated amygdala responsivity to threat-related stimuli as well as deficient top-down modulation of amygdala responses by specific cortical regions, including the pregenual anterior cingulate cortex, subcallosal cortex, and hippocampus.

The investigators propose to investigate the pathophysiology of several specific anxiety disorders, Posttraumatic Stress Disorder (PTSD), Panic Disorder (PD), and Specific Phobia(SP), by using cognitive activation paradigms and magnetic resonance imaging (MRI) to probe the function and structure of implicated amygdalo-cortical circuitry.

DETAILED DESCRIPTION:
All candidates for this project will undergo a comprehensive clinical assessment by an investigator trained to administer these instruments. At the MGH fMRI Center in Charlestown or at the Neuroimaging Center at McLean Hospital in Belmont, MA; each subject will undergo a single MRI session lasting approximately 2 hours. After the scanning session, subjects may be asked to make judgments about the facial expressions or the words that were presented.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age
* Right-handed (Edinburgh Inventory - Oldfield 1971)
* SCID diagnosis consistent with group designation:

Current PTSD (PTSD group; none current or past (NC and TENC group); Current SP (must be to small animal phobia, SP group); Current PD (PD group)

* To be matched for age, gender, and years of education, as well as self-identified race/ethnicity.
* For female subjects, stage of menstrual cycle will be ascertained by history (see appendix), and dates of fMRI acquisition will be scheduled to prevent systematic differences between groups with respect to this variable.

Exclusion Criteria:

* Neurologic or medical condition that would interfere with study procedures or confound results, ascertained by history.
* History of seizure or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion)
* History of exclusionary Axis I psychiatric diagnosis (other than as specified); i.e., history of substance use disorder, psychotic disorder, bipolar disorder, tic disorder, or eating disorder. Note that comorbid current major depressive disorder will be allowed in up to one half of each study group. This will enable inclusion of this common comorbidity, but also enable a definitive assessment of whether or not the presence of this comorbid diagnosis is driving any observed significant between group differences.
* Use of psychotropic medication within 4 weeks prior to study (within 6 weeks for fluoxetine, or other long-lived compounds; within one year for neuroleptics).
* Pregnancy (to be ruled out by urine ß-HCG).
* Metallic implants or devices contraindicating magnetic resonance imaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Boston metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
amygdala activation during Masked Affect Task | measured once at fMRI session

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Rauch, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Rosso IM, Makris N, Britton JC, Price LM, Gold AL, Zai D, Bruyere J, Deckersbach T, Killgore WD, Rauch SL. Anxiety sensitivity correlates with two indices of right anterior insula structure in specific animal phobia. Depress Anxiety. 2010 Dec;27(12):1104-10. doi: 10.1002/da.20765. PMID 21132846
- [Result] Killgore WD, Britton JC, Price LM, Gold AL, Deckersbach T, Rauch SL. Neural correlates of anxiety sensitivity during masked presentation of affective faces. Depress Anxiety. 2011 Mar;28(3):243-9. doi: 10.1002/da.20788. Epub 2011 Feb 9. PMID 21308886
- [Result] Britton JC, Gold AL, Deckersbach T, Rauch SL. Functional MRI study of specific animal phobia using an event-related emotional counting stroop paradigm. Depress Anxiety. 2009;26(9):796-805. doi: 10.1002/da.20569. PMID 19434621